CLINICAL TRIAL: NCT05022355
Title: The Comparison of the Effects of Scapulothoracic Arthrodesis Surgery Versus Usual Care on Balance and Gait Parameters in Patients With Fascioscapulohumeral Dystrophy: One-Blind Study
Brief Title: Examination of Operative Approach in pwFSHD (Patient With Facioscapulohumeral Muscular Dystrophy)
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysenur Erekdag, BSc, Istanbul University - Cerrahpasa
Other Study IDs: 38981562-900-
Record Dates: First submitted 2021-08-21; First posted 2021-08-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Facio-Scapulo-Humeral Dystrophy
Keywords: scapulotorasic arthrodesis; balance; gait; evaluation; usual care
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- scapulothoracic arthrodesis: Individuals diagnosed with FSHD who have undergone unilateral or bilateral surgery who meet the inclusion criteria.
  application of determined outcome scales on patients
- non-operative: Participants diagnosed with FSHD who have not undergone any surgery, who meet the inclusion criteria.
  application of determined outcome scales on patients

SUMMARY:
Facioscapulohumeral Muscular Dystrophy (FSHD) is one of the most common forms of muscular dystrophy, characterized by pronounced skeletal novelistic weakness and with a broad spectrum of diseases. It is a hereditary disease seen in 3-5/100,000 of society, usually starting with weakness in the facial and shoulder muscles and progressing to the trunk, pelvis and leg muscles, giving symptoms in the twenties. In FSHD, which shows slow progression and can lead to loss of ambulation ability in about 20% of patients, patients may have difficulty performing activities above shoulder level with the influence of the periscapular area.

Skeletal muscle weakness leads to posture and balance disorders, and postural instability is a common problem in patients with FSHD. Weakness of the trunk and lower limb muscles found in more than half of patients causes problems with postural balance and walking. The calf, iliopsoas, and gluteus maximus muscles together form the main determinants of walking speed in healthy people, where kalf muscles are known to contribute the most. Individuals with FSHD have been reported to have decreased speed, step length, and step frequency compared to healthy controls. Impaired upper body control can compromise the maintenance of dynamic stability. In patient with FSHD the effects of muscle tone, motor coordination, loss of joint range of motion and muscle weakness on posture, balance control and gait are observed more clearly.

The aim of the study was to compare the effects of scapular management treatments on balance and gait in FSHD patients.

H0: There is no difference in balance and walking parameters of patients with FSHD who have had scapulothoracic arthrodesis surgery and have not undergone surgery.

H1: There is a difference in balance and walking parameters of patients with FSHD who have had scapulothoracic arthrodesis surgery and have not undergone surgery.

DETAILED DESCRIPTION:
Voluntary patients who have been diagnosed with FSHD will be included in the study. Signed voluntary consent will be obtained from participants. Participants will be divided into two groups. One group will include patients who have undergone scapulothoracic arthrodesis surgery, while the other group will include patients who have not undergone surgery. Both groups will undergo some outcome measures to assess their balance and walking.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years
* Score between 0,5 and 3,5 according to CSS (clinical severity rating)
* Score between 3 and 5 according to FAS (functional ambulation scale)
* Being included in the surgical group the patient has undergone unilateral or bilateral scapulothoracic arthrodesis surgery

Exclusion Criteria:

* Presence of lower extremity orthopedic problems/problems that can cause balance and walking problems
* Presence of any other upper limb orthopedic problems/problems and surgery
* Having undergone Spinal fusion surgery
* Presence of additional neurological problems/problems
* Having a level of visual and auditory problems that will prevent communication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients diagnosed with FSHD and undergoing scapulothoracic arthrodesis or non-operating
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2022-08-16 (Actual)

PRIMARY OUTCOMES:
10 meter walking test | once at baseline of study
  during the test, the patient is asked to walk at a normal walking speed at a distance of 10 meters determined before the test. The time it has traveled the specified distance is recorded. It is a long-term performance test used for dynamic balance assessment.
Gait Analyzer | once at baseline of study
  It is a smartphone-based application for analyzing walking parameters in real time. It can measure walking speed, step time, step length, cadence and symmetry.

SECONDARY OUTCOMES:
Berg Balance Scale | once at baseline of study
  It is a scale containing 14 instructions and a score of 0-4 is given by observing the patient's performance for each instruction. 0 points are given in cases where the patient cannot perform the activity at all, while 4 points are given when the patient completes the activity independently. The highest score is 56 and 0-20 points indicate balance disorder, 21-40 points indicate an acceptable balance, 41-56 points indicate the presence of a good balance. It takes between 10 and 20 minutes to complete the scale.
Disabilities of the arm, shoulder and hand (DASH) | once at baseline of study
  It is a 30-item questionnaire that examines the patient's ability to perform certain upper limb activities. This survey is a self-report questionnaire in which patients can assess difficulty and intervention in daily life on a Likert scale of 5 points.
30 seconds sit up test | once at baseline of study
  It is a test that evaluates the patient's sit-up activity, lower limb strength and dynamic balance. A 30-second period is initiated when the patient cuts the contact of his pelvis from the chair in which he is sitting. He is constantly asked to sit on the chair and get up from there within 30 seconds. It is scored by counting how many repetitions the patient applies this command within 30 seconds.
2-minute walk test | once at baseline of study
  it is recommended that the area where the test will be performed should be a corridor with a length of 30 meters, a flat and hard floor. It is necessary to determine the starting and ending points of the field to be tested. The patient is asked to walk the maximum distance he can walk within 2 minutes by standing at the starting point. When it expires, the distance it travels is recorded.
Single leg stance test | once at baseline of study
  It is used to evaluate static posture and balance control. The patient must stand unaided on one leg from the moment the other foot leaves the ground until the foot touches the ground again or the arms are separated from the hips.
Timed up and go test | once at baseline of study
  The Test is a measure of dynamic equilibrium. It requires individuals to get up from a chair, walk 3 feet, turn and sit. The time from the moment the individual lifts the pelvis from the chair until he or she returns with the pelvis in the chair is recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ipek Yeldan, PhD, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Fecek C, Emmady PD. Facioscapulohumeral Muscular Dystrophy. 2023 Jun 26. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK559028/ PMID 32644454
- [Background] Rijken NH, van Engelen BG, Weerdesteyn V, Geurts AC. Clinical Functional Capacity Testing in Patients With Facioscapulohumeral Muscular Dystrophy: Construct Validity and Interrater Reliability of Antigravity Tests. Arch Phys Med Rehabil. 2015 Dec;96(12):2201-6. doi: 10.1016/j.apmr.2015.08.429. Epub 2015 Sep 9. PMID 26363336
- [Background] Tawil R, Van Der Maarel SM. Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2006 Jul;34(1):1-15. doi: 10.1002/mus.20522. PMID 16508966
- [Background] Bayram S, Kendirci AS, Karalar S, Durmus Tekce H, Parman FY, Akgul T, Durmaz H. Correlations between radiographic spinopelvic parameters and health-related quality of life: A prospective evaluation of 37 patients with facioscapulohumeral muscular dystrophy. Clin Neurol Neurosurg. 2020 Nov;198:106137. doi: 10.1016/j.clineuro.2020.106137. Epub 2020 Aug 5. PMID 32791439
- [Background] Padua L, Aprile I, Frusciante R, Iannaccone E, Rossi M, Renna R, Messina S, Frasca G, Ricci E. Quality of life and pain in patients with facioscapulohumeral muscular dystrophy. Muscle Nerve. 2009 Aug;40(2):200-5. doi: 10.1002/mus.21308. PMID 19609906
- [Background] Kang PB, Morrison L, Iannaccone ST, Graham RJ, Bonnemann CG, Rutkowski A, Hornyak J, Wang CH, North K, Oskoui M, Getchius TS, Cox JA, Hagen EE, Gronseth G, Griggs RC; Guideline Development Subcommittee of the American Academy of Neurology and the Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Evidence-based guideline summary: evaluation, diagnosis, and management of congenital muscular dystrophy: Report of the Guideline Development Subcommittee of the American Academy of Neurology and the Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Neurology. 2015 Mar 31;84(13):1369-78. doi: 10.1212/WNL.0000000000001416. PMID 25825463
- [Background] Tawil R, Kissel JT, Heatwole C, Pandya S, Gronseth G, Benatar M; Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology; Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Evidence-based guideline summary: Evaluation, diagnosis, and management of facioscapulohumeral muscular dystrophy: Report of the Guideline Development, Dissemination, and Implementation Subcommittee of the American Academy of Neurology and the Practice Issues Review Panel of the American Association of Neuromuscular & Electrodiagnostic Medicine. Neurology. 2015 Jul 28;85(4):357-64. doi: 10.1212/WNL.0000000000001783. PMID 26215877
- [Background] Le Hanneur M, Saint-Cast Y. Long-term results of Letournel scapulothoracic fusion in facioscapulohumeral muscular dystrophy: A retrospective study of eight cases. Orthop Traumatol Surg Res. 2017 May;103(3):421-425. doi: 10.1016/j.otsr.2016.12.012. Epub 2017 Jan 31. PMID 28159680
- [Background] Kord D, Liu E, Horner NS, Athwal GS, Khan M, Alolabi B. Outcomes of scapulothoracic fusion in facioscapulohumeral muscular dystrophy: A systematic review. Shoulder Elbow. 2020 Apr;12(2):75-90. doi: 10.1177/1758573219866195. Epub 2019 Aug 14. PMID 32313557
- [Background] Statland JM, Tawil R. Risk of functional impairment in Facioscapulohumeral muscular dystrophy. Muscle Nerve. 2014 Apr;49(4):520-7. doi: 10.1002/mus.23949. Epub 2014 Feb 10. PMID 23873337
- [Background] Iosa M, Mazza C, Pecoraro F, Aprile I, Ricci E, Cappozzo A. Control of the upper body movements during level walking in patients with facioscapulohumeral dystrophy. Gait Posture. 2010 Jan;31(1):68-72. doi: 10.1016/j.gaitpost.2009.08.247. Epub 2009 Sep 25. PMID 19782569
- [Background] Rijken NH, van der Kooi EL, Hendriks JC, van Asseldonk RJ, Padberg GW, Geurts AC, van Engelen BG. Skeletal muscle imaging in facioscapulohumeral muscular dystrophy, pattern and asymmetry of individual muscle involvement. Neuromuscul Disord. 2014 Dec;24(12):1087-96. doi: 10.1016/j.nmd.2014.05.012. Epub 2014 Jun 26. PMID 25176503
- [Background] Aprile I, Padua L, Iosa M, Gilardi A, Bordieri C, Frusciante R, Russo G, Erra C, De Santis F, Ricci E. Balance and walking in facioscapulohumeral muscular dystrophy: multiperspective assessment. Eur J Phys Rehabil Med. 2012 Sep;48(3):393-402. Epub 2012 Jun 20. PMID 22713540
- [Background] Rijken NH, van Engelen BG, de Rooy JW, Weerdesteyn V, Geurts AC. Gait propulsion in patients with facioscapulohumeral muscular dystrophy and ankle plantarflexor weakness. Gait Posture. 2015 Feb;41(2):476-81. doi: 10.1016/j.gaitpost.2014.11.013. Epub 2014 Dec 2. PMID 25687333